CLINICAL TRIAL: NCT04965571
Title: Clinical Features and Outcome of Wilson's Disease With Generalized Epilepsy in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: WD-seizures
Record Dates: First submitted 2021-07-05; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Wilson Disease; Generalized Epilepsy
Keywords: Chinese; clinical features; generalized epilepsy; outcome; Wilson's disease
MeSH Terms: conditions — Hepatolenticular Degeneration; Epilepsy, Generalized | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- WD-seizures: Chinese WD patients with generalized epilepsy
  Interventions: Genetic: genetic test

INTERVENTIONS:
Genetic: genetic test — Sanger sequencing and multiplex ligation-dependent probe amplification (MLPA)

SUMMARY:
Generalized epilepsy is rarely reported in patients with Wilson disease (WD) and lacks experience in clinical practice. We aim to provide better experience for the diagnosis and treatment for WD patients with epilepsy in the future.

DETAILED DESCRIPTION:
A retrospective study was performed in 13 Chinese WD patients with generalized epilepsy. Each patient was diagnosed with WD by clinical evaluation and genetic screening. Patients were given small doses of antiepileptic drugs (AEDs), followed by copper-chelation therapy when the seizures stabilized. Clinical manifestations, brain imaging changes, and treatment and outcome after a long-term follow-up were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Each patient was diagnosed with WD by clinical evaluation and genetic screening and had ever experienced generalized epilepsy

Exclusion Criteria:

* Not WD & without generalized epilepsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each patient was diagnosed with WD by clinical evaluation and genetic screening. Patients were given small doses of antiepileptic drugs (AEDs), followed by copper-chelation therapy when the seizures stabilized.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment stop seizures attacks | 12 month
  After standard treatment, the patients would stop attacks and get improved.

SECONDARY OUTCOMES:
Number of participants with treatment have improved brain MRI | 12 month
  After standard treatment, the abnormalities of brain MRI would get better in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided